CLINICAL TRIAL: NCT00001119
Title: A Study of the Effects of Combination Antiretroviral Therapy in Acute HIV-1 Infection With an Emphasis on Immunological Responses
Brief Title: Effects on the Immune System of Anti-HIV Drugs in Patients Recently Infected With HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Purpose: Treatment
Other Study IDs: AIEDRP AI-02-001
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2011-03-02 (Estimated); Status verified 2005-01

CONDITIONS: HIV Infections
Keywords: Immunity, Cellular; Drug Therapy, Combination; HIV Protease Inhibitors; Antibody Formation; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load; Tetanus Toxoid; Case-Control Studies; Hepatitis B Surface Antigens; Acute Infection
MeSH Terms: conditions — HIV Infections; Tetanus; Hepatitis B | interventions — Tetanus Toxoid; Indinavir; lamivudine, zidovudine drug combination; Ritonavir; abacavir; amprenavir; efavirenz; Hepatitis B Vaccines; Lamivudine; Zidovudine

INTERVENTIONS:
Biological: Tetanus Toxoid Vaccine
Drug: Indinavir sulfate
Drug: Lamivudine/Zidovudine
Drug: Ritonavir
Drug: Abacavir sulfate
Drug: Amprenavir
Drug: Efavirenz
Biological: Hepatitis B Vaccine (Recombinant)
Drug: Lamivudine
Drug: Zidovudine

SUMMARY:
The purpose of this study is to find out whether these powerful combinations of anti-HIV drugs are safe and effective for use in patients in the early stages of HIV infection and to find out how patients' immune systems react to HIV and anti-HIV drugs.

Doctors generally treat patients in the early stages of HIV infection with the same anti-HIV drugs taken by patients who have had HIV for a long time. These drugs lower the level of HIV in the blood. However, doctors do not know whether patients who take anti-HIV drugs in the early stages of HIV infection actually live longer or have fewer AIDS-related diseases. This study will help doctors answer these questions. In the main study, doctors will look at how 2 different anti-HIV drug combinations affect the immune system. In the 2 substudies, doctors will look at how the body reacts to the hepatitis B vaccine and the tetanus vaccine. These substudies may help doctors learn how HIV-infected patients respond to new infections.

DETAILED DESCRIPTION:
Current treatment guidelines recommend combination ART for acute primary HIV-1 infection. However, it is not known whether ART given during acute infection delays progression to AIDS or improves survival rates. Preliminary studies suggest ART given early in HIV infection not only reduces viral load but also restricts CD4+ cell loss, delays the development of opportunistic infections, and preserves T-helper cells and naive T cells. The immunologic basis of these protective effects has not been characterized thoroughly. This protocol assesses ART's effects on immune responses in early HIV infection through a variety of cellular, humoral, and virologic assays, including 2 substudies. The substudies focus on antibody responses to neoantigen immunization (hepatitis B and tetanus). Primary endpoint analysis occurs at Week 72, but patients may be followed for long-term outcomes.

In the main study, patients with HIV-1 infection of less than 120 days are given the option of taking a potent ART combination of abacavir (ABC), efavirenz (EFV), indinavir (IDV), and lamivudine (3TC) for 96 weeks. [AS PER AMENDMENT 9/15/00: Patients choose either Regimen 1: ABC, 3TC, IDV, and ritonavir (RTV) or Regimen 2: ABC, 3TC, and EFV.] Patients who decline treatment provide a concurrent, non-randomized comparison group. These patients may choose to be considered for study treatment at any time or to start antiretrovirals provided through another source. [AS PER AMENDMENT 9/15/00: If a patient who initially does not start therapy subsequently starts antiretroviral therapy provided by the study (within the 120-day limit), the visit schedule is re-set.] During the treatment period, all patients undergo regular physical exams and blood tests to characterize T cells, viral resistance, antibody responses, and other markers. Patients presenting within 30 days of HIV-1 infection undergo leukapheresis (where available) prior to starting ART. At Month 12, these patients and all untreated patients undergo leukapheresis to assess the proportion of latently infected CD4+ T cells. In addition, all patients in the main study and patients in 2 comparison groups (Cohorts A and B) participate in 1 of 2 substudies of antibody responses to neoantigen. Volunteers are recruited to 2 cohorts to serve as controls. Cohort A volunteers have established HIV-1 infection. Cohort B volunteers are HIV-1 seronegative but at high risk for HIV. In the first substudy, hepatitis B-seronegative patients from the main study and from Cohorts A and B receive hepatitis B vaccine at Weeks 40, 44, and 64 and undergo humoral and cellular response assessments at Week 68. In the second substudy, patients from the main study and from Cohorts A and B who did not qualify for the hepatitis B vaccination undergo intramuscular vaccination with tetanus toxoid at Week 64 and immune responses are assessed at Week 68. Volunteers in Cohorts A and B receive no anti-HIV medication as part of these substudies.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for the main study if they:

* Became infected with HIV within the last 120 days.
* Are at least age 16 and have written consent of a parent or guardian if under 18.
* Are willing to practice abstinence or use barrier methods of birth control, such as condoms.
* Are available for at least 72 weeks.
* Patients may be eligible for 1 of the 2 substudies if they:
* Are at least age 16 and have written consent of a parent or guardian if under 18.
* Have had HIV infection for more than 1 year and have a CD4 cell count greater than 500 cells/mm3, or do not have HIV infection but are at risk of getting HIV because of their lifestyle, such as sexual activity or injection drug use.
* Have never had hepatitis B infection or a hepatitis B vaccine and they are available for 28 weeks (hepatitis B vaccine substudy only).
* Have not received a tetanus shot in the past 5 years, have never had an allergic reaction to a tetanus shot, and are available for 8 weeks (tetanus shot substudy only).

Exclusion Criteria

Patients will not be eligible for the main study if they:

* Have taken anti-HIV drugs for more than 7 days for the treatment of HIV. However, anti-HIV drugs taken to help prevent HIV are acceptable.
* Have certain types of cancer.
* Are receiving an experimental treatment.
* Are pregnant or breast-feeding.
* Are allergic to study drugs.
* Have taken certain medications that may interfere with the study.
* Patients will not be eligible for 1 of the 2 substudies if they:
* Are receiving an experimental treatment.
* Are pregnant or breast-feeding.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 288
Dates: Start 1999-10; Primary Completion 2004-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Corey, Study Chair
Locations (12):
- United States (11):
  - San Francisco Dept of Hlth / AIDS Office, San Francisco, California
  - Univ of Illinois Chicago / Howard Brown Hlth Ctr, Chicago, Illinois
  - Fenway Community Health Ctr / HIVNET, Boston, Massachusetts
  - Univ of Minnesota, Minneapolis, Minnesota
  - New York Univ Med Ctr, New York, New York
  - Bronx-Lebanon Hosp Ctr, The Bronx, New York
  - Univ of Cincinnati, Cincinnati, Ohio
  - Mem Hosp of Rhode Island, Pawtucket, Rhode Island
  - Seattle HIVNET, Seattle, Washington
  - Univ of Washington, Seattle, Washington
  - Fred Hutchinson Cancer Research Ctr, Seattle, Washington
- Saint Vincent's Hosp Med Centre, Darlinghurst, Australia

REFERENCES:
- [Result] Stekler J, Maenza J, Stevens C, Holte S, Malhotra U, McElrath MJ, Corey L, Collier AC. Abacavir hypersensitivity reaction in primary HIV infection. AIDS. 2006 Jun 12;20(9):1269-74. doi: 10.1097/01.aids.0000232234.19006.a2. PMID 16816555